CLINICAL TRIAL: NCT00282620
Title: The Adjuvant Magnesium Trial (AdMag): Assessment if the Impact of Oral Magnesium on ICD Firing and Quality of Life
Brief Title: Magnesium to Reduce Implantable Cardioverter Defibrillator (ICD) Shocks and Improve Patient's Quality of Life.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hartford Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KLUG001817HE
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-03

CONDITIONS: Arrhythmia; Quality of Life; Hypomagnesemia
Keywords: Implantable Cardioverter Defibrillator; Magnesium; Electrocardiogram; Ventricular Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

INTERVENTIONS:
Drug: Magnesium L-lactate

SUMMARY:
This study is being conducted to see if magnesium can reduce the number of shocks patients with ICDs experience and to see if magnesium supplementation improves patients quality of life.

DETAILED DESCRIPTION:
Not all ICD shocks are for ventricular arrhythmias. Some patients receive shocks when they have arrhythmias in the atria (top chambers of the heart). These are called inapproriate shocks, but the pain is similar to the pain patients feel with an appropriate shock (a shock for a ventricular arrhythmia). This study is being conducted to determine if taking magnesium can reduce the number of shocks patients with ICDs experience and to see if magnesium supplementation improves patients quality of life. Magnesium's impact of the electrocardiogram (ECG) and intracellular magnesium concentrations will also be studied.

Comparison: Magnesium compared to placebo in patients with ICDs to evaluate the number of ICD shocks and patient perceived quality of life.

ELIGIBILITY:
Inclusion Criteria:newly implanted ICD or recent ICD shock (within 6 months) -

Exclusion Criteria:inability to swallow, a non-cardiac disease with a survival prognosis of less than 12 months, hypermagnesemia, a creatinine clearance less than 30mL/min, lactic acidosis or systemic acidosis syndrome, or previous intolerance to magnesium L-lactate.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2006-01; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative occurrence of ICD shocks and patient perceived quality of life at baseline, 3,6,9, and 12 months

SECONDARY OUTCOMES:
Change in QTc interval in the total population and the subgroup receiving class III antiarrhythmics at baseline, 3, 6, 9, 12 months.
Intracellular magnesium concentrations at baseline, 3 and 12 months
Incidence of supraventricular arrhythmias, ventricular arrhythmias, and sinus tachycardias at baseline, 3,6,9,12 months.
Ventricular fibrillation cycle length and the variability in VFCL at baseline, 3,6,9,12 months
Adverse events at basline, 3,6,9,12 months. Total Hospital Costs and Cost-effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kluger, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States